CLINICAL TRIAL: NCT03405233
Title: Role of Double Cuffed PTFE Arteriovenous Grafts in Enhancing Long-term Patency in Hemodialysis Patients: a Randomized Controlled Trial
Brief Title: Role of Double Cuffed PTFE Arteriovenous Grafts in Enhancing Long-term Patency in Hemodialysis Patients (Extended Poly Tetra Fluoro Ethylene)
Acronym: ePTFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Elshafie, Assistant Lecturer of vascular surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.18.01.6.R1
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease
Keywords: ESRD; ePTFE; neointemal hyperplasia
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the patients do not know which group will they belong the duplex operator will not know the details of operative data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Double vein cuff PTFE graft both at the inflow and outflow ends
  Interventions: Procedure: Double vein cuffed ePTFE graft both at the inflow and outflow ends
- Group B (Active Comparator): Single vein cuffed PTFE graft at the outflow end
  Interventions: Procedure: single vein cuffed eTFE graft both at the inflow and outflow ends
- Group C (Active Comparator): PTFE graft without vein cuff will be used
  Interventions: Procedure: ePTFE graft without any cuff

INTERVENTIONS:
Procedure: Double vein cuffed ePTFE graft both at the inflow and outflow ends — Vein cuff is obtained from a segment of one of the arm veins (cephalic or basilica) after incising it longitudinally and wrapped around both ends of PTFE Graft
  Arms: Group A
Procedure: single vein cuffed eTFE graft both at the inflow and outflow ends — Vein cuff is obtained from a segment of one of the arm veins (cephalic or basilica) after incising it longitudinally and wrapped around the venous end of PTFE Graft
  Arms: Group B
Procedure: ePTFE graft without any cuff — anastmosis between arterial and venous side usinf non cuffed ePTFE graft
  Arms: Group C

SUMMARY:
this randomized controlled trial will compare the double vein cuffed synthetic arteriovenous graft to the single vein cuffed synthetic and the non cuffed synthetic as regard to long-term patency of each modality

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) arises from many heterogeneous disease pathways that alter the function and structure of the kidney irreversibly, over months or years.End-stage renal disease (ESRD) arises from many heterogeneous disease pathways that alter the function and structure of the kidney irreversibly, over months or years. Haemodialysis (HD) is a lifeline therapy for patients with ESRD. A proportion of hemodialysis patients exhaust all options for permanent vascular access (fistula or graft) in both upper extremities.ePTFE grafts are easily subjected to graft outflow tract intimal hyperplasia, which may lead to graft outlet stenosis and graft thrombosis after a certain period of usage. The commonest cause of PTFE graft failure is intimal hyperplasia (IH) at the venous anastomoses. our study aims to evaluate the influence of double cuffed ePTFE grafts with autologous vein cuffs on the long-term patency of dialysis access, and compare the clinical patency and the complications occurring with the usage of the double cuffed graft to that with standard non cuffed grafts in chronic renal hemodialysis therapy.

this randomized controlled trial will compare the double vein cuffed synthetic arteriovenous graft to the single vein cuffed synthetic and the non cuffed synthetic as regard to long term patency of each modality

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end stage renal diseases and GFR less than 30
2. By clinical examination in ability to palpate distal or proximal upper limb veins 3. By duplex examination the diameter of cephalic or basilic veins are less than 3 mm or reported to be incompressible 4. Patients with previous history of failed attempts of autogenous vein creation 5. Patients with border line cephalic or basilica vein (3mm) and on intraoperative the vein diameter appears to be unsuitable (less than 3 mm).

Exclusion Criteria:

1. All patients with palpable suitable forearm or arm veins
2. Patients with baseline blood pressure less than 110/70
3. Brachial artery of diameter less than 4 mm
4. Patients with ligated brachial artery
5. Patients with history of central vein stenosis
6. Patients with immunodeficiency states

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
primary patency | 2 years for each patient after the operation
  comparing primary patency between the double cuffed, single cuffed and non cuffed ePTFE graft primary patency means how long will the graft be patent after the first intervention

SECONDARY OUTCOMES:
secondary patency | 2 years after restoration of patency
  comparing secondary patency between the double cuffed, single cuffed and non cuffed ePTFE graft secondary patency means how long will the graft be patent after thormobectomy to a thrombosed graft

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Delta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng C, Tempel D, van Haperen R, van der Baan A, Grosveld F, Daemen MJ, Krams R, de Crom R. Atherosclerotic lesion size and vulnerability are determined by patterns of fluid shear stress. Circulation. 2006 Jun 13;113(23):2744-53. doi: 10.1161/CIRCULATIONAHA.105.590018. Epub 2006 Jun 5. PMID 16754802
- [Background] Ghonemy TA, Farag SE, Soliman SA, El-okely A, El-hendy Y. Epidemiology and risk factors of chronic kidney disease in the El-Sharkia Governorate, Egypt. Saudi J Kidney Dis Transpl. 2016 Jan;27(1):111-7. doi: 10.4103/1319-2442.174137. PMID 26787576
- [Background] Ong S, Barker-Finkel J, Allon M. Long-term outcomes of arteriovenous thigh grafts in hemodialysis patients: a comparison with tunneled dialysis catheters. Clin J Am Soc Nephrol. 2013 May;8(5):804-9. doi: 10.2215/CJN.09240912. Epub 2013 Jan 31. PMID 23371958
- [Background] Tsoulfas G, Hertl M, Ko DS, Elias N, Delmonico FL, Romano L, Fernandes I, Schoenfeld D, Kawai T. Long-term outcome of a cuffed expanded PTFE graft for hemodialysis vascular access. World J Surg. 2008 Aug;32(8):1827-31. doi: 10.1007/s00268-008-9514-z. PMID 18343971